CLINICAL TRIAL: NCT04489420
Title: A Phase I Study of Human Placental Hematopoietic Stem Cell Derived Natural Killer Cells (CYNK-001) in Adults With Recurrent Glioblastoma Multiforme (GBM)
Brief Title: Natural Killer Cell (CYNK-001) IV Infusion or IT Administration in Adults With Recurrent GBM
Acronym: CYNK001GBM01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision.
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYNK001-GBM-001
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Astrocytoma, Grade IV; Giant Cell Glioblastoma; Glioblastoma Multiforme; Cyclophosphamide; Immunosuppressive Agents; Immunologic Factors; Physiological Effects of Drugs; Molecular Mechanisms of Pharmacological Action; Antiviral Agents; Anti-infective Agents; Analgesics, Non-narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents
Keywords: CYNK-001; Glioblastoma Multiforme; Grade IV Astrocytoma; allogeneic; allogeneic stem cell; GBM; cell therapy; Cyclophosphamide; recurrent GBM; recurrent Glioblastoma Multiforme; primary and secondary recurrent GBM; NK cells; natural killer cells
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: 2 modalities Systemic vs Intratumoral. For systemic experimental: Cyclophosphamide at Day -3 followed by CYNK-001. On Days 0, 7, and 14. Experimental IntraTumoral, Ommaya placement surgery 7 days prior to CYNK-001 administrations at Days 0, 7 and 14
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous IV ( Recurrent and Surgical ) GBM (Experimental): Cohort 1A ( recurrent GBM) will receive CYNK-001 at a dose of 1.2 x 10^9 cells intravenous ( IV) on Days 0, 7, and 14 and will include up to 6 subjects. The subjects will be followed for a 42 day DLT period from the initial CYNK-001 infusion (or 28 days after the last dose). No other treatment interventions are planned between the last day of CYNK-001. In the event of DLTs, Cohort 1C ( recurrent GBM dose-De escalation) will receive CYNK-001 at a dose of 600 x 10^6 cells (IV) on Days 0, 7, 14, and will include up to 6 subjects who will be followed for a 42-day DLT period from the initial CYNK-001 infusion (or 28 days after the last dose. Cohort 1B (surgical cohort) will receive CYNK-001 at the maximum safe dose (MSD) (either 1.2x10^9 cells or 600x10^6 cells) (IV) at Days 0, 7, 14, and will include up to 6 subjects. The tumor resection surgery will be performed after the last CYNK-001 infusion during the DLT period.
  Interventions: Biological: CYNK001-IV
- Intratumoral IT ( Recurrent and Surgical ) GBM) (Experimental): The cohort 2A or cohort 2C (recurrent GBM) IT route of administration can be started only after the safety results were acceptable from the completion of cohort 1A or Cohort 1C (IV route of administration). The Treatment Period for the IT cohorts will begin with having the Ommaya catheter placement per institutional policy, which is planned to occur within one week prior to the CYNK-001 administration on Day 0. Cohort 2A will be treated with CYNK-001 IT at 200 x 10^6 ± 50 x 10^6 cells IT on Day 0, 7 and 14 includes up to 6 recurrent GBM subjects Cohort 2C ( dose de-escalation) will be treated with CYNK-001 200 x 106 ± 50 x 106 cells IT on Day 0, and Day 7 ( only two days dosing) and include up to 6 recurrent GBM subjects. Cohort 2B ( the surgical IT cohort) will be treated with CYNK-001 at the maximum safe dose ( MSD) (either 200 x 10^6 ± 50 x 10^6 cells on Days 0, 7 and 14 or at 200 x 10^6 ±50x10^6 cells on Days 0 and 7) and include up to 6 surgical GBM subjects
  Interventions: Biological: CYNK001-IT

INTERVENTIONS:
Biological: CYNK001-IV — Planned Starting dose dor IV 1.2x10^9 cells/dose
  Other Names: CYNK-001 dose level 1 for IV
  Arms: Intravenous IV ( Recurrent and Surgical ) GBM
Biological: CYNK001-IT — Planned starting dose for IT 200 x10^6 +/- 50 x10^6 cells dose
  Other Names: CYNK-001 dose level 2 for IT
  Arms: Intratumoral IT ( Recurrent and Surgical ) GBM)

SUMMARY:
This study will find the maximum safe dose (MSD) or maximum tolerated dose (MTD) of CYNK-001 which are NK cells derived from human placental CD34+ cells and culture-expanded. CYNK-001 cells will be given after lymphodepleting chemotherapy for the systemic cohort (IV) (intravenous). The intratumoral cohort (IT) will not be giving lymphodepletion. The safety of this treatment will be evaluated, and researchers want to learn if NK cells will help in treating recurrent glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed glioblastoma multiforme (GBM) and are at first or second relapse.
2. ≥ 18 years of age
3. Have measurable disease of at least one solitary lesion with a dimension between 1 cm and 5 cm according to RANO
4. Karnofsky performance status (KPS) ≥ 60
5. Adequate organ function defined by laboratory values as follows: Creatinine < 140 µmol/L (1.6 mg/dL); if borderline, the creatinine clearance ≥40 mL/min, Bilirubin < 20% above the upper limit of normal, AST and ALT ≤ 2.5 the upper limit of normal.
6. Absolute Neutrophil count baseline (ANC) ≥1500 cells/uL, Hemoglobin baseline ≥ 9.0 g/dL and Platelets baseline ≥ 100,000 cells/uL prior to the start of study treatment.
7. Female of childbearing potential (FCBP) must not be pregnant and agree to not becoming pregnant for at least 42 days following the start of the treatment.
8. Patients with HIV/AIDs are eligible if they have not had an opportunistic infection within the past 12 months
9. Patients with chronic HBV infection or patients with current or a history of HCV infection are allowed if:

   1. have an HBV viral load below the limit of quantification and be on viral suppressive therapy
   2. have current HCV infection, they should be on concurrent HCV treatment and the HCV viral load must be below the limit of quantification
   3. have a history of HCV infection should have completed curative antiviral treatment and require HCV viral load below the limit of quantification

Exclusion Criteria:

1. Had prior radiation therapy within 12 weeks of screening MRI unless there is unequivocal histological confirmation of tumor progression
2. Subjects on growth factors therapy with less than 4 weeks washout period (for short-acting growth factors, such as G-CSF, GM-CSF 5-day wash-out for longer-acting factors (such as Neulasta) 10 days
3. Radiotherapy, chemotherapy, or other investigational agents within 4 weeks
4. Prior cellular or gene therapy at any time
5. Clinical or laboratory signs for immunodeficiency or under immunosuppressive medication or steroids greater than15 mg prednisone or equivalent per day
6. History of malignancy, other than GBM, unless the subject has been free of disease for > 3 years from the date of signing the ICF. Exceptions include the following noninvasive malignancies: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
7. Active autoimmune disease other than controlled connective tissue disorder or those who are not on active therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants who experienced a Dose-Limiting Toxicity (DLT) | Day 42
  Defined as the maximum dose safely administered intravenously or Intratumoral for the treatment of patients with GBM.
Adverse Events (AEs) | 1 year
  Defined as the number and Severity of Adverse Events

SECONDARY OUTCOMES:
Overall Response Rate | 1 year
  Defined as the proportion of subjects with best overall response of either complete response (CR) or partial response (PR)
Duration of Response Rate | 1year
  Defined as duration from first observation of partial response (PR) or better to the date of disease progression per RANO criteria
Progression-free survival | 1year
  Defined as date of the first CYNK-001 infusion to the date of disease progression per RANO Response Criteria or death (regardless of cause of death), whichever comes first
Time to porgression | 1year
  Defined as the date of the first CYNK-001 infusion to the date of disease progression per RANO Response Criteria, with deaths from causes other than progression censored
Overall Survival | 1year
  Defined as the date of the first CYNK-001 infusion to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Koppisetti, MD, Study Director — Celularity inc.
Locations (1):
- The Univeristy of Texas MD ANderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided